CLINICAL TRIAL: NCT06889597
Title: The Effects of Virtual and Mixed Reality Exergaming on Mood and Executive Functioning During Micro Breaks at Work: A Randomized Crossover Trial
Brief Title: Effects of VR and MR Exergaming on Mood and Executive Function During Workplace Microbreaks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Abdullah Kayhan, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 06032025-05-118
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Exergame; Active Video Games (AVG); Mood State; Executive Function (Cognition)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR EXERGAME (Experimental): Participants will engage in a Virtual Reality (VR)-based exergame session using the PowerBeatsVR application. The session will include rhythm-based exercises, such as punching targets and dodging obstacles, aimed at promoting physical activity during a short break in the workplace.
  Interventions: Other: Experimental
- MR EXERGAME (Experimental): Participants will engage in a Mixed Reality (MR)-based exergame session using the PowerBeatsVR application in MR mode. This condition allows participants to interact with virtual elements while maintaining awareness of their physical surroundings.
  Interventions: Other: Experimental
- REST (No Intervention): Participants will remain seated in a quiet room for the same duration as the VR and MR sessions. During this time, they will be asked to rest without engaging in any physical activity. Talking, using mobile devices, or interacting with others will not be allowed to ensure a consistent resting condition across participants.

INTERVENTIONS:
Other: Experimental — Virtual Reality Exergame (VR) Participants will engage in a 5-minute fully immersive Virtual Reality (VR) exergame session using the PowerBeatsVR application. This intervention takes place in a virtual environment where participants perform rhythm-based physical activities such as punching targets and dodging obstacles. The VR session isolates participants from their real-world surroundings, offering a highly immersive experience designed to promote physical activity and assess its physiological and psychological effects.
  Other Names: VR EXERGAME
  Arms: MR EXERGAME
Other: Experimental — Mixed Reality Exergame (MR) Participants will engage in a 5-minute Mixed Reality (MR) exergame session using PowerBeatsVR in MR mode. Unlike VR, this intervention integrates virtual elements into the real-world environment, allowing participants to maintain awareness of their physical surroundings while interacting with digital content. This hybrid experience reduces the risk of cybersickness while providing a practical approach for workplace settings.
  Other Names: MR EXERGAME
  Arms: VR EXERGAME

SUMMARY:
This study aims to evaluate the effects of virtual reality (VR) and mixed reality (MR) exergaming interventions during workplace microbreaks on mood and executive functions. A crossover experimental design will be implemented with desk-based administrative employees. Participants will be randomly assigned to three conditions: VR exergaming, MR exergaming, and passive rest. Executive functions will be assessed using the PEBL Victoria Stroop Test, and mood state will be evaluated with the Positive Affect Subscale of PANAS (PA-PANAS). Secondary measures include heart rate, perceived exertion, and exercise adherence intention.The study will address the following research questions:

How do VR and MR exergames influence executive functions compared to passive rest? How do VR and MR exergames affect mood states in workers compared to passive rest? How do VR and MR exergames compare in terms of heart rate response and perceived exertion during workplace microbreaks? How do VR and MR exergames impact exercise enjoyment and the intention to continue exergaming?

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* No regular physical exercise in the last three months (less than three days per week, less than 30 minutes per session)
* No prior experience with VR/MR technologies
* No history of neurological or cardiovascular disorders
* No epilepsy, vertigo, or inner ear conditions
* No use of medications affecting the central nervous system
* Low or moderate physical activity levels, as assessed by the International Physical Activity Questionnaire (IPAQ)
* Cleared for physical activity based on the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* High physical activity levels as indicated by the IPAQ
* Not meeting the safety criteria for physical activity according to the PAR-Q
* Individuals experiencing dizziness, nausea, or discomfort while using VR/MR
* Vision impairments that prevent the use of VR/MR headsets
* Pregnant individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Executive Functions | Baseline and immediately post-intervention (within 5 minutes after the session
  Executive functions will be assessed using the PEBL Victoria Stroop Test. This test evaluates cognitive control, reaction time, and error rates in different experimental conditions. To eliminate learning effects, each participant will complete two practice trials before the experimental session. The test consists of three phases (1. Neutral words (words without color conflict), 2. Congruent words (words where the meaning matches the text color), 3.Incongruent words (words where the meaning differs from the text color).
  Participants will be instructed to identify the color of the word as quickly and accurately as possible. Reaction times (in milliseconds) and error rates will be recorded.
Mood State | Baseline and immediately post-intervention (within 5 minutes after the session)
  Participants' mood states will be assessed using the Positive Affect subscale of the Positive and Negative Affect Schedule (PANAS). PANAS is a widely used self-report instrument designed to measure two distinct dimensions of affective states: Positive Affect (PA) and Negative Affect (NA). However, in this study, only the PA subscale will be utilized. This decision is based on the study's focus on the short-term affective benefits of VR and MR exercise, as physical activity is predominantly linked to improvements in positive emotions rather than significant reductions in negative affect. Additionally, since negative emotions may not exhibit substantial changes in a single-session exercise context, analyzing only positive affect provides a clearer understanding of the intervention's psychological benefits.

SECONDARY OUTCOMES:
Heart Rate | Baseline and during intervention
  Heart rate will be measured using a Polar H10 chest strap sensor at two time points: pre-exercise and during the session. All HR data will be recorded in real time via the Polar Flow application. The HR measurements will be used to assess the physiological load of the exercise and compare differences across conditions.
Perceived Exertion | Baseline and immediately post-intervention (within 5 minutes after the session)
  Subjective physical exertion will be evaluated using the Borg Rating of Perceived Exertion (RPE) Scale (6-20) before and after each session. This scale measures subjective physical effort perception and is widely used for assessing exercise intensity.
Intention to Continue | Immediately post-intervention (within 5 minutes after the session)
  Participants' intention to engage in VR and MR-based exercise in the future will be measured using a 7-point Likert scale (1 = Not at all likely, 7 = Definitely will repeat). Higher scores indicate a stronger intention to continue using VR/MR-based exercise programs in the future. This outcome will help determine the long-term engagement potential of immersive exercise formats.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Konyaalti, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No